CLINICAL TRIAL: NCT02833740
Title: Field Testing of a Set of Simplified Mid-upper Arm Circumference Classification Devices ("Click-MUAC") for Use by Mothers and Caregivers to Screen for Acute Malnutrition in Young Children at Community Level, in Isiolo County, Kenya
Brief Title: Comparing Performance of Simplified Mid-Upper Arm Circumference Devices ("Click-MUACs") to Detect Acute Malnutrition
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Action Contre la Faim (Other)
Collaborators: Tampere University (Other); Brixton Health (Unknown); Humanitarian Innovation Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: USG5A
Record Dates: First submitted 2016-05-12; First posted 2016-07-14 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Malnutrition
Keywords: Mid-Upper Arm Circumference (MUAC); Mother MUAC; Community screening for acute malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Click-MUAC & regular MUAC tape screening (Other): Each child will have nutritional status classified 11 times:
  * 3 times with each of the 3 Click-MUAC prototypes by the mother/caregiver
  * 1 time with a regular MUAC tape by the mother/caregiver
  * 3 times with each of the 3 Click-MUAC prototypes by the case-finding/programme staff
  * 1 time with a regular MUAC tape by the case-finding/programme staff
  * 3 times with a regular MUAC tape by the data collection team ("gold standard")
  Interventions: Device: Click-MUAC prototype & regular MUAC tape

INTERVENTIONS:
Device: Click-MUAC prototype & regular MUAC tape — Screening of children using Click-MUAC and regular MUAC tape

SUMMARY:
The Click-Mid-Upper Arm Circumference study aims to describe and compare the performance of a set of three simplified mid-upper arm circumference classification devices ("Click-MUAC") for use by mothers and caregivers to screen for acute malnutrition in young children. The study will be conducted in Isiolo County, Kenya. The study builds on the recent approach of training mothers to screen for acute malnutrition in their own children (mother MUAC approach).

The primary aim of the study is to describe and compare the performance of a set of three prototype Click-MUAC devices against a gold standard of classification, in terms of measures of agreement (sensitivity, specificity, accuracy, Cohen's Kappa, Youden's J) for the classification (diagnosis) of acute malnutrition. A secondary aim of the study is to determine the difference in agreement with the gold standard classification amongst mothers/caregivers using a Click-MUAC prototype versus mothers/caregivers using a regular MUAC tape. The hypothesis of the study is that at least one of the Click-MUAC prototypes is equal to the gold standard of classification in terms of measures of agreement for the classification of acute malnutrition. A secondary hypothesis of the study is that agreement with the gold standard classification is better amongst mothers/caregivers using a Click-MUAC prototype compared to mothers/caregivers using a regular MUAC tape. The outcomes of the study will be used to decide on whether production of a Click-MUAC device is desirable and, if this is the case, to select a design based on the performance of the prototype devices and the stated preferences of intended users.

DETAILED DESCRIPTION:
The study will be a non-randomised, non-blinded, clinical diagnostic trial describing and comparing performance that will be conducted in two phases: (i) calibration of the devices, (ii) testing of Click-MUAC prototypes against "gold standard" classification.

The study will take place at designated health facilities within Isiolo County that already have an IMAM programme running. The investigators expect that the health facilities with the highest number of acute malnutrition admissions will be selected as study sites in order to be able to test the prototypes on a large number of attending Severe Acute Malnutrition (SAM)/Moderate Acute Malnutrition (MAM) children.

The first phase of work will concentrate on the calibration of Click-MUAC prototypes. The performance of the Click-MUAC prototypes with regard to accuracy of classification will be assessed in children with a measured MUAC at or close to the 115 mm and 125 mm case-defining thresholds. This phase of work is required as prior testing of the Click-MUAC prototypes will only have been performed on semi-rigid testing tubes.

The second phase of work will test the Click-MUAC prototypes. Three sets of measurements/classifications will be taken during the Click-MUAC testing trial: (i) Mother/caregiver MUAC classification performed by the mother/primary caregiver on their own child, using each of the three Click-MUAC prototypes and a regular MUAC tape; (ii) IMAM staff MUAC classification performed by the Integrated Management of Acute malnutrition (IMAM) staff on the same child, using each of the three Click-MUAC prototypes and a regular MUAC tape; (iii) Gold standard MUAC measurement performed by the study coordinator and/or data collection team members trained in the measurement of MUAC and selected for their accuracy (i.e. against the study supervisor) and precision of measurement, following a validation exercise using the Habicht method, on the same child. In addition, mothers/caregivers and IMAM staff will also be asked to state their preference of Click-MUAC prototype and asked to give reasons for their preference.

The Click-MUAC devices are screening/diagnostic devices. Appropriate measures of agreement between the different measurer groups (mothers/primary caregivers, IMAM staff, gold standard) can be calculated from two-by-two contingency tables. The following appropriate measures of agreement will be calculated from these tables: sensitivity, specificity, accuracy, Cohen' s Kappa, Younden's J. The analysis (i.e. two-by-two contingency table and estimation of appropriate measures of agreement) will be performed for each prototype Click-MUAC device. A discordancy analysis will also be performed. The aim of the discordancy analysis is to describe misclassifications in terms of the range, interquartile range, and median MUAC at each type of discordancy. This analysis provides further calibration information that may inform design changes that avoid/minimize gross misclassifications and to minimize the frequency of errors made at or close to class boundaries.

ELIGIBILITY:
Inclusion Criteria:

* Child 6-59 months with MUAC < 115 mm presenting at health facility for treatment of acute malnutrition or identified at paediatric outpatient clinic.
* Child 6-59 months with MUAC < 115 mm currently enrolled in IMAM programme
* Child 6-59 months with MUAC between 115 mm and 125 mm presenting at health facility for treatment of acute malnutrition or identified at paediatric outpatient clinic.
* Child 6-59 months with MUAC between 115 mm and 125 mm currently enrolled in IMAM programme.
* Child 6-59 months with MUAC ≥ 125 mm identified at paediatric outpatient clinic.

AND informed consent of mother / caregiver

Exclusion Criteria:

* Child < 6 months or >59 months.
* Child with physical handicap preventing mid-upper arm circumference measurement.
* Child requiring immediate and urgent medical attention for medical complications.
* Child with mid-upper arm skin lesions (e.g. scabies, impetigo, ringworm).
* Bilateral pitting oedema.
* Caregiver consent not given.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 345 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Youden's J | Immediate (i.e. this measure can be calculated immediately upon data collection). The measure will be collected throughout study implementation for up to 3 months, for completion as planned for October 2016.
  Youden's J is a chance-corrected measure of agreement that can be interpreted as the probability of making an informed decision using a given method of ascertaining case-status. The measure is estimated as:
  J = Sensitivity + Specificity - 1
  Sensitivity is defined as the ability of the Click-MUAC device to correctly detect patients who do have the condition (i.e. either severe wasting or moderate wasting or any wasting). The measure is mathematically defined as: sensitivity = a/(a+b) where a= true positive and b= false negative
  Specificity is defined as the ability of the Click-MUAC device to correctly detect patients who do not have the condition (i.e. either severe wasting or moderate wasting or any wasting). The measure is mathematically defined as specificity= d/(c+d) where d=true negative and c=false positive

SECONDARY OUTCOMES:
Accuracy | Immediate (i.e. this measure can be calculated immediately upon data collection). The measure will be collected throughout study implementation for up to 3 months, for completion as planned for October 2016.
  The term "accuracy" best applies to agreement between true case status (from the gold standard measurement procedure) and classification by mothers or program staff.
  The measure is mathematically defined as accuracy= (a+d)/(a+b+c+d) where a= true positive, b= false negative, c=false positive and d=true negative
Cohen's Kappa | Immediate (i.e. this measure can be calculated immediately upon data collection). The measure will be collected throughout study implementation for up to three months, for completion as planned for October 2016.
  Cohen's Kappa is defined mathematically as:
  Cohen's Kappa= (p_o-p_e)/(1-p_e )
  The term p_o is observed agreement (calculated from the two-by-two contingency table) and the term p_e is expected agreement (also calculated from the two-by-two contingency table). Cohen's Kappa can be used with square contingency tables larger than the two-by-two case. The measure is useful for evaluating a Click-Mid-Upper Arm Circumference (MUAC) device for more than two classes (e.g. severe wasting, moderate wasting, no wasting).

CONTACTS AND LOCATIONS:
Overall Officials: Angeline E Folliet-Grant, Principal Investigator — Action Against Hunger | ACF-USA
Locations (1):
- Isiolo County Health Facilities implementing integrated management of acute malnutrition (IMAM), Isiolo, Isiolo County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grant A, Njiru J, Okoth E, Awino I, Briend A, Murage S, Abdirahman S, Myatt M. Comparing performance of mothers using simplified mid-upper arm circumference (MUAC) classification devices with an improved MUAC insertion tape in Isiolo County, Kenya. Arch Public Health. 2018 Feb 22;76:11. doi: 10.1186/s13690-018-0260-x. eCollection 2018. PMID 29484177